CLINICAL TRIAL: NCT05890534
Title: Pycnogenol® in People With Post-COVID-19 Condition: a Quadruple-blind, Randomized, Placebo-controlled Trial
Brief Title: Pycnogenol® in Post-COVID-19 Condition
Acronym: PYCNOVID
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-01967
Record Dates: First submitted 2023-06-05; First posted 2023-06-06 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Post COVID-19 Condition; Long COVID
Keywords: COVID-19; post COVID symptoms; Pycnogenol®
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — pycnogenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data analyst is also masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pycnogenol® (Experimental): People with post COVID-19 condition randomly allocated to the Pycnogenol® arm will take 4 capsules of Pycnogenol® per day (4x50mg capsules, 200mg total) over a period of 12 weeks.
  Interventions: Drug: Pycnogenol®
- Placebo (Placebo Comparator): People with post COVID-19 condition randomly allocated to the Placebo arm will take 4 capsules of Placebo per day (4x50mg capsules, 200mg total) over a period of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pycnogenol® — Single center, quadruple blind randomized controlled trial comparing Pycnogenol® versus Placebo.
  Arms: Pycnogenol®
Drug: Placebo — Single center, quadruple blind randomized controlled trial comparing Pycnogenol® versus Placebo.
  Arms: Placebo

SUMMARY:
To determine the effect of Pycnogenol® versus placebo on patient-reported health status in people with post COVID-19 condition.

DETAILED DESCRIPTION:
The primary aim of this 12-week quadruple blind, single-center randomized controlled trial is to determine the effect of Pycnogenol® (200mg daily) versus placebo on patient-reported health status (EQ-Visual Analogue Scale) in people with post COVID-19 condition. Secondary outcomes include symptoms, fatigue, cognitive function, health-related quality of life, functional exercise capacity and blood biomarkers of inflammation, endothelial function and oxidative stress.

Pycnogenol® is a licensed pine tree bark extract (Pinus pinaster ssp. atlantica) and primarly used for the treatment of venous disorders. Various studies reported beneficial effects in other conditions such as diabetes, metabolic syndrome and cardiovascular disorders. Pycnogenol® exerts antioxidative, anti-inflammatory and antiproliferative effects and has been shown to improve vascular endothelial function. Pycnogenol® may have potential to improve the health status of people suffering from post COVID-19 condition.

This trial lasts for 12 weeks. Participants are invited to visit the study center four times: screening visit, baseline visit, follow-up 1 visit (6 weeks after baseline visit), follow-up 2 visit (12 weeks after baseline visit).

In a substudy using baseline data, the investigators plan to study associations between objectively measured physical activity, severity of post COVID-19 condition, symptom burden and severity (e.g., fatigue, dyspnoea), functional exercise capacity, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection confirmed by positive PCR or rapid antigen test for professional use or written medical report
* Post-COVID condition (WHO definition), i.e., ≥ 3 months after SARS-CoV2 infection and ongoing or recurring symptoms for at least 2 months that cannot be explained by alternative diagnosis
* Symptoms include fatigue and / or cognitive impairment ("brain fog") and / or dyspnea and / or post-exertional malaise
* Willing to participate and having signed informed consent
* Sufficient language and cognitive skills
* Ability to participate in study visits
* No foreseeable change in medication

Exclusion Criteria:

* Severe comorbidities such as liver or renal failure, advanced COPD or pulmonary fibrosis requiring > 5L oxygen/min at rest, active malignancy, advanced heart failure, cardio-vascular events within the previous 24 weeks (such as unstable coronary artery disease, coronary revascularization, myocardial infarction, stroke, transient ischemic attack, critical limb ischemia, pulmonary embolism, deep vein thrombosis), uncontrolled severe hypertension, uncontrolled diabetes uncontrolled autoimmune or inflammatory disease (the responsible study physician will decide each case on an individual basis)
* Acute respiratory or other infections (postpone baseline visit until resolved)
* Clinical diagnosis of a psychiatric disease (e.g., depression, anxiety disorder, schizophrenia) that is untreated and/or unstable (the responsible study physician will decide each case on an individual basis)
* COVID-19 vaccination less than 4 weeks prior to the baseline visit (i.e., first or second dose of a two-dose vaccination regimen, first dose of a single dose vaccination regimen, booster) or during study participation (booster shot will be offered at screening visit, wait time until baseline visit 4 weeks)
* Known intolerance of the study drug
* Regular intake of Pycnogenol®
* Pregnancy or lactating. For women and transgender individuals of childbearing age, who can anamnestically not exclude a pregnancy, are offered a pregnancy test during the study visits.
* Being enrolled in another interventional study that may interfere with the current study (the responsible study physician will decide each case on an individual basis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Health status (EQ-VAS) | Change from baseline to 12 weeks
  EQ-Visual Analogue Scale (EQ-VAS also known as "Feeling thermometer") assessed daily over 7 consecutive days prior to the baseline and at the end of the follow-up 2 visit (i.e., study end after 12 weeks). The scale ranges from 0-100 with 0 representing worst health status and 100 representing best health status.

SECONDARY OUTCOMES:
Post COVID-19 symptoms | Change from baseline to 12 weeks
  Symptoms (present/not present) and symptom severity (5- point Likert scale: 1=not bad at all, 2=mild, 3=moderate, 4=severe, 5=very severe) will be assessed using a self-administered online questionnaire. Symptoms will also be recorded in a paper diary and completed on a weekly basis.
Fatigue | Change from baseline to 12 weeks
  Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F). 13-item questionnaire with a 7-day recall period assessed at baseline and after 12 weeks. The level of fatigue is measured on a 5-point Likert scale (4 = not at all fatigued to 0 = very much fatigued). Individual item scores are summed, with lower scores indicating more severe fatigue.
Dyspnea | Change from baseline to 12 weeks
  Symptom domain of the Chronic Respiratory Questionnaire (CRQ) assessed at baseline and after 12 weeks. The questionnaire contains 5 questions; 7-point Likert-type scale ranging from 1 (most severe dyspnea) to 7 (no dyspnea).
Cognitive function | Change from baseline to 12 weeks
  Montreal Cognitive Assessment (MoCA) assessed at baseline and after 12 weeks. The cut-off score < 26 for cognitive impairment will be used in this study.
Anxiety and depression | Change from baseline to 12 weeks
  Hospital, Anxiety and Depression Scale (HADS) assessed at baseline and after 12 weeks. Symptoms of depression and anxiety (14 questions, 4-point Likert-type scale).
Health-related quality of life (EQ-5D-5L) | Change from baseline to 12 weeks
  The EQ-5D-5L assesses the 5 dimensions mobility, self-care, usual activities, pain/discomfort, anxiety/depression. The EQ-5D-5L scores each dimension on five levels of severity ranging from 1 = "no problems" to 5 = "extreme problems. The instrument will be used at baseline and after 12 weeks.
Functional exercise capacity | Change from baseline to 12 weeks
  A 30 second Sit-to-Stand (STS) will be performed at baseline and after 12 weeks. The number of repetitions that the participant completes the full sit-to-stand movement on a chair during 30 seconds. A familiarisation test will be done at the screening visit to rule out potential learning effects.
Physical activity | Change from baseline to 12 weeks
  Physical activity measured with an accelerometer (ActiGraph wGT3X-BT, Pensacola, FL, USA), which is worn at the right hip over 8 consecutive days prior to the baseline and 12 week study visit. Number of daily steps and time spent in different intensity domains (min per day) will be analysed.
Soluble Thrombomodulin (sTM) | Change from baseline to 12 weeks
  Blood biomarker of endothelial health measured with Enzyme-linked Immunosorbent Assay (ELISA) or Luminex (bead-based immunoassay) at baseline and after 12 weeks.
von Willebrand Factor antigen (VWF:Ag) | Change from baseline to 12 weeks
  Blood biomarker of endothelial health measured with Enzyme-linked Immunosorbent Assay (ELISA) or Luminex (bead-based immunoassay) at baseline and after 12 weeks.
Syndecan-1 | Change from baseline to 12 weeks
  Blood biomarker of endothelial health measured with Enzyme-linked Immunosorbent Assay (ELISA) or Luminex (bead-based immunoassay) at baseline and after 12 weeks.
Circulating Cascular Cell Adhesion Molecule-1 (sVCAM 1) | Change from baseline to 12 weeks
  Blood biomarker of endothelial health measured with Enzyme-linked Immunosorbent Assay (ELISA) or Luminex (bead-based immunoassay) at baseline and after 12 weeks.
C-reative protein (CRP) | Change from baseline to 12 weeks
  Marker of inflammation (serum) measured at baseline and after 12 weeks by a certified laboratory (Analytica, Zurich, Switzerland).
Interleukine 6 (IL 6) | Change from baseline to 12 weeks
  Marker of inflammation measured with Enzyme-linked Immunosorbent Assay (ELISA) or Luminex (bead-based immunoassay) at baseline and after 12 weeks.
sCD40L | Change from baseline to 12 weeks
  Marker of coagulation and platelet function measured with Enzyme-linked Immunosorbent Assay (ELISA) or Luminex (bead-based immunoassay) at baseline and after 12 weeks.
sP selectin | Change from baseline to 12 weeks
  Adhesion molecule measured with Enzyme-linked Immunosorbent Assay (ELISA) or Luminex (bead-based immunoassay) at baseline and after 12 weeks.
D-Dimer | Change from baseline to 12 weeks
  Marker of coagulation and platelet function measured in citrate blood at baseline and after 12 weeks by certified laboratory (Analytica, Zurich, Switzerland).
Activated partial thromboplastin time (aPTT) | Change from baseline to 12 weeks
  Marker of coagulation and platelet function measured in citrate blood at baseline and after 12 weeks by certified laboratory (Analytica, Zurich, Switzerland).
International normalized ratio (INR) blood test | Change from baseline to 12 weeks
  Marker of coagulation and platelet function measured in citrate blood at baseline and after 12 weeks by certified laboratory (Analytica, Zurich, Switzerland).
Total antioxidant capacity (TAC) | Change from baseline to 12 weeks
  Marker of oxidative stress measured in blood plasma at baseline and after 12 weeks. TAC will be measured using the well-established Ferric Reduction Capability of Plasma (FRAP) method using a commercially available kit.
Aspartate aminotransferase (ASAT) | Change from baseline to 12 weeks
  Marker of liver function measured in blood serum at baseline and after 12 weeks by a certified laboratory (Analytica, Zurich, Switzerland).
Alanine aminotransferase (ALAT) | Change from baseline to 12 weeks
  Livery enzyme measured in blood serum at baseline and after 12 weeks by a certified laboratory (Analytica, Zurich, Switzerland).
Gamma glutamyltransferase (γ-GT) | Change from baseline to 12 weeks
  Livery enzyme measured in blood serum at baseline and after 12 weeks by a certified laboratory (Analytica, Zurich, Switzerland).
Creatinine | Change from baseline to 12 weeks
  Creatinine including clearance measured in blood serum at baseline and after 12 weeks by a certified laboratory (Analytica, Zurich, Switzerland).

OTHER OUTCOMES:
Adherence to study products | Baseline to 12 weeks
  Adherence to study products (Pycnogenol® and Placebo) will be evaluated during the two follow-up visits (6 and 12 weeks after baseline visit) and the two follow-up phone calls using a standardized assessment form. The number of capsules returned at the study visits will be counted and entered into the database.
Post-exertional malaise | Baseline to 12 weeks
  Post-exertional malaise is a frequent symptom in post COVID-19 condition. Study visits and measurements may pose a burden for the participants. At each visit, starting with the baseline visit, participants will be asked whether they experienced a worsening of their symptoms within 3 days after the last study visit (i.e., after 12 weeks). A self-administered questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jahn S Fehr, Prof., MD, Study Director — University of Zurich, EBPI, Department of Public & Global Health; Alexia Anagnostopoulos, MD, Principal Investigator — University of Zurich, EBPI, Department of Public & Global Health
Locations (1):
- University of Zurich, Epidemiology, Biostatistics and Prevention Institute, Department of Public & Global Health, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radtke T, Kunzi L, Kopp J, Rasi M, Braun J, Zens KD, Winter B, Anagnostopoulos A, Puhan MA, Fehr JS. Effects of Pycnogenol(R) in people with post-COVID-19 condition (PYCNOVID): study protocol for a single-center, placebo controlled, quadruple-blind, randomized trial. Trials. 2024 Jun 15;25(1):385. doi: 10.1186/s13063-024-08187-6. PMID 38879571